CLINICAL TRIAL: NCT03204617
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Safety, Tolerability and Immunogenicity Study of Candidate HIV-1 Vaccines DNA.HTI, MVA.HTI and ChAdOx1.HTI in Early Treated HIV-1 Positive Individuals
Brief Title: Safety and Immunogenicity Study of DNA.HTI, MVA.HTI and ChAdOx1.HTI in HIV-1-positive Patients (AELIX-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aelix Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AELIX-002
Record Dates: First submitted 2017-06-13; First posted 2017-07-02 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: HIV
Keywords: HIV infection; First in Human; Therapeutic Vaccines; HTI; HIV reservoir
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind: two or more parties are unaware of the intervention assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DDDMM + CCM (Experimental): DNA.HTI 0.5mL at weeks 0, 4 and 8 + MVA.HTI 0.5mL at weeks 12 and 20. At least 24 weeks since second MVA.HTI administration (week 20), administration of ChAdOx1.HTI 0.5mL at weeks 0 and 12 + MVA.HTI 0.5mL at week 24.
  Interventions: Biological: DNA.HTI 0.5mL at weeks 0, 4 and 8 + MVA.HTI 0.5mL at weeks 12 and 20 (DDDMM); Biological: At least 24 weeks since DDDMM, ChAdOx1.HTI 0.5mL at weeks 0 and 12 + MVA.HTI 0.5mL at week 24 (CCM)
- Placebo (Placebo Comparator): 0.9% sterile normal saline solution at weeks 0, 4, 8, 12 and 20. At least 24 weeks since fifth placebo administration, administration of 0.9% sterile normal saline solution at weeks 0, 12 and 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: DNA.HTI 0.5mL at weeks 0, 4 and 8 + MVA.HTI 0.5mL at weeks 12 and 20 (DDDMM) — Vaccine DNA.HTI 0.5mL at weeks 0, 4 and 8 + Vaccine MVA.HTI 0.5mL at weeks 12 and 20 (DDDMM).
  Other Names: N/H
  Arms: DDDMM + CCM
Biological: At least 24 weeks since DDDMM, ChAdOx1.HTI 0.5mL at weeks 0 and 12 + MVA.HTI 0.5mL at week 24 (CCM) — At least 24 weeks since second MVA.HTI administration (week 20), administration of ChAdOx1.HTI 0.5mL at weeks 0 and 12 + MVA.HTI 0.5mL at week 24.
  Other Names: N/H
  Arms: DDDMM + CCM
Drug: Placebo — 0.9% sterile normal saline solution at weeks 0, 4, 8, 12 and 20. At least 24 weeks since the fifth Placebo administration, 0.9% sterile normal saline solution at weeks 0, 12 and 24
  Other Names: N/H
  Arms: Placebo

SUMMARY:
The AELIX-002 study aims to evaluate the safety and the immunogenicity of an heterologous prime-boost regimen with DNA.HTI, MVA.HTI and ChAdOx1.HTI in early diagnosed and treated HIV-1 positive individuals, males and females,18-60 years of age.

DETAILED DESCRIPTION:
AELIX Therapeutics has developed a novel immunogen, which was designed to be used as a a therapeutic HIV vaccine that could help HIV infected individuals to control viral replication in the absence of antiretroviral treatment. HIVACAT T cell immunogen (HTI) is a novel T cell immunogen covering the most vulnerable regions of HIV. The encoding DNA sequence that has been inserted in various vaccine vectors, including viral and non-viral vectors. Administration of the HTI immunogen is implemented through a heterologous prime-boost approach. The aim of the sequential administration of the therapeutic vaccines is to achieve a so-called "functional cure," in which HIV-infected participants can control viral replication in the absence of ART.

The AELIX-002 Phase I study will evaluate the safety and immunogenicity of an heterologous regime with DNA.HTI, MVA.HTI and ChAdOx1.HTI in HIV-1 positive participants on suppressive antiretroviral treatment who started Combination Antiretroviral Therapy (cART) within the first 6 months of confirmed HIV-1 acquisition. In Phase A, participants were randomized to receive active vaccine or placebo in a double blinded fashion. There was a sentinel group of three participants; two received active vaccine and one received placebo (0.9% normal saline). During the sentinel phase of the study only one participant was enrolled per day. Two weeks later and in the absence of any related SAE or ≥ Grade 3 adverse event lasting >72h after vaccination in any of the 3 sentinel participants, six individuals in the remaining cohort were enrolled (in blocks of 3 patients per day) and the final six participants one week later, also in blocks of 3 participants per day. On each vaccination day, 2 participants received active IMP and 1 received placebo (2:1).

After the first 15 participants (3 sentinel and 12 non-sentinel) have reached week 22 visit and a favourable report from the Safety Monitoring Committee has been released, transition to Phase B was performed to include 30 participants (Group 3). Participants were recruited sequentially and without following blocks of pre-defined number of vaccines and placebos per immunization day.

At week 32, all participants were invited to participate in an extension sub-study (Roll-over Phase) to assess long-term safety, tolerability and immunogenicity of DNA.HTI and MVA.HTI administrations until start of Phase C. There were no interventions during this extension Roll over Phase.

After a favourable SMC report, transition to Phase C occurred. During Roll-over Phase participants in Phase A/B were offered to participate in Phase C. Participants who received active treatment (DDDMM) in Phase A/B will continue to receive active treatment (CCM) in Phase C, while participants who received placebo in Phase A/B will continue to receive placebo (PPP). Treatment allocation remained blind. Eight weeks after the third MVA.HTI/placebo administration, all participants will undergo an Analytical Treatment Interruption (ATI) of up to 24 weeks of duration. At visit Phase C week 56 (end-of-ATI visit), or before according to pre-specified criteria, cART will be resumed, and participants will be followed during a safety period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV-1 infection
2. On combined antiretroviral treatment (defined as ≥ 3 antiretroviral drugs) initiated within 6 months of estimated time of HIV-1 acquisition.
3. Willing and able to be adherent to their cART regimen for the duration of the study.
4. Optimal virological suppression for at least 1 year defined as maintained pVL below the limit of detection (based on current available assays, 20, 40 or 50 copies/ml) allowing for isolated blips.
5. Being on the same cART regimen for at least 4 weeks at screening visit.
6. Nadir CD4 count ≥ 200 cells per mm3. Isolated lower counts at the moment of acute HIV-1 infection will be allowed only if appropriate immune recovery was followed after cART initiation (as is criteria 7).
7. Stable CD4 counts ≥ 400 cells per mm^3 for the last 6 months at screening visit.
8. Availability of stored biological sample (including PBMC and plasma) before any cART initiation.
9. Aged at least 18 years on the day of screening and no greater than 60 years on the day of the first vaccination.
10. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
11. In the opinion of the principal investigator or designee, the patient has understood the information provided and capable of giving written informed consent.
12. If heterosexually active female; using an effective method of contraception (hormonal contraception, intra-uterine device (IUD), or anatomical sterility in self or partner) from 14 days prior to the first vaccination until at least 12 weeks after the last vaccination; all female volunteers must be willing to undergo urine pregnancy tests at time points specified in the Schedule of Procedures.
13. If heterosexually active male; willing to use an effective method of contraception (anatomical sterility in self) or agree on the use of an effective method of contraception by his partner (hormonal contraception, intra-uterine device (IUD), or anatomical sterility) from the day of the first vaccination until 12 weeks after the last vaccination.
14. Willing to accept blood draws and collect stool at time points specified in the Schedule of Procedures.
15. Willing to forgo donating blood during the study.

Exclusion Criteria:

1. Pregnancy or lactating.
2. Presence of resistance drug mutations in a pre-cART genotype.
3. Reported periods of suboptimal adherence to cART.
4. History of past antiretroviral treatment interruptions longer than 2 weeks.
5. Participation in another clinical trial within 12 weeks of study entry (at screening visit).
6. Any AIDS-defining disease or progression of HIV-related disease.
7. History of autoimmune disease.
8. History or clinical manifestations of any physical or psychiatric disorder which could impair the subject's ability to complete the study.
9. Receipt of approved vaccines within 2 weeks of study entry and along the duration of the trial.
10. History of anaphylaxis or severe adverse reaction to vaccines.
11. Previous immunisation with any experimental immunogens.
12. Receipt of blood products within 6 months of study entry.
13. Treatment for cancer or lymphoproliferative disease within 1 year of study entry.
14. Any other current or prior therapy which, in the opinion of the investigators, would make the individual unsuitable for the study or influence the results of the study.
15. Current or recent use (within last 3 months) of interferon or systemic corticosteroids or other immunosuppressive agents (use on inhaled steroids for asthma or topic steroids for localized skin conditions are permitted).
16. Any laboratory abnormalities including:

    Haematology
    * Haemoglobin < 10.0 g/dl
    * Absolute Neutrophil Count (ANC) ≤ 1,000 /mm3
    * Absolute Lymphocyte Count (ALC) ≤ 600 /mm3
    * Platelets ≤100,000 /mm3, ≥ 550,000 /mm3

    Biochemistry
    * Creatinine > 1.3 x ULN
    * Aspartate aminotransferase (AST) > 2.5 x ULN
    * Alanine aminotransferase (ALT) > 2.5 x ULN

    Microbiology
    * Positive for hepatitis B surface antigen,
    * Positive for hepatitis C antibody, unless confirmed clearance of HCV infection (spontaneous or following treatment)
    * Positive serology indicating active syphilis requiring treatment
17. Complete refusal to cART interruption

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Proportion of participants that develop Grade 3 or 4 local reactions | From first DNA.HTI/Placebo administration to week 32 and from first ChAdOx1.HTI/Placebo administration to week 32
  Grade 3 or 4 local reactions as assessed by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events
Proportion of participants that develop Grade 3 or 4 systemic reactions | From first DNA.HTI/Placebo administration to week 32 and from first ChAdOx1.HTI/Placebo administration to week 32
  Grade 3 or 4 systemic reactions as assessed by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events

SECONDARY OUTCOMES:
Proportion of participants that develop T cell responses to HTI-encoded regions | From first DNA.HTI/Placebo administration to week 32 and from first ChAdOx1.HTI/Placebo administration to week 32
  Proportion of patients that develop T cell responses to HTI-encoded regions as determined by IFN-γ ELISPOT assay in vaccine and placebo recipients
Breadth of total vaccine induced HIV-specific responses | From first DNA.HTI/Placebo administration to week 32 and from first ChAdOx1.HTI/Placebo administration to week 32
  Breadth of total vaccine induced HIV-specific responses measured IFN-γ ELISPOT in vaccine and placebo recipients
Magnitude of total vaccine induced HIV-specific responses | From first DNA.HTI/Placebo administration to week 32 and from first ChAdOx1.HTI/Placebo administration to week 32
  Magnitude of total vaccine induced HIV-specific responses measured IFN-γ ELISPOT in vaccine and placebo recipients
Percentage of participants with viral remission, defined as plasma viral load (pVL) <50 copies/mL 12 and 24 weeks after start of Analytical Treatment Interruption (ATI) | From ATI start (visit Phase C week 32) to weeks 12 and 24 after ATI start (visits Phase C week 44 and week 56).
  Percentage of participants with viral remission, defined as plasma viral load (pVL) <50 copies/mL 12 and 24 weeks after start of ATI
Percentage of participants with pVL <2,000 copies/mL at 12 and 24 weeks after start of ATI | From ATI start (visit Phase C week 32) to weeks 12 and 24 after ATI start (visits Phase C week 44 and week 56).
  Percentage of participants with pVL <2,000 copies/mL at 12 and 24 weeks after start of ATI
Time to viral detection, defined as the time from ATI start (visit Phase C week 32) to first occurrence of detectable pVL (>50 copies/mL) | From ATI start (visit Phase C week 32) to first occurrence of detectable pVL (>50 copies/mL) up to week 56
  Time to viral detection, defined as the time from ATI start (visit Phase C week 32) to first occurrence of detectable pVL (>50 copies/mL).
Time to viral rebound, defined as the time from ATI start (visit Phase C week 32) to first occurrence of pVL >10,000 copies/mL. | From ATI start (visit Phase C week 32) to first occurrence of pVL >10,000 copies/mL up to week 56
  Time to viral rebound, defined as the time from ATI start (visit Phase C week 32) to first occurrence of pVL >10,000 copies/mL.
Percentage of participants who remain off cART at 12 and 24 weeks after ATI (visits Phase C week 44 and week 56). | From ATI start (visit Phase C week 32) to weeks 12 and 24 after ATI start (visits Phase C week 44 and week 56).
  Percentage of participants who remain off cART at 12 and 24 weeks after ATI (visits Phase C week 44 and week 56).
Time off cART, defined as time to cART resumption since ATI start (visit Phase C week 32). | From ATI start (visit Phase C week 32) to cART resumption through study completion, up to week 68
  Time off cART, defined as time to cART resumption since ATI start (visit Phase C week 32).
Proportion of participants who develop symptoms compatible with acute retroviral syndrome (ARS) during ATI. | From ATI start (visit Phase C week 32) to cART resumption up to week 56
  Proportion of participants who develop symptoms compatible with acute retroviral syndrome (ARS) during ATI.
Proportion of participants who develop new mutations not present in the pre-cART genotype conferring clinically-significant resistance to antiretroviral drugs (out of the individuals not reaching viral re-suppression 12 weeks after cART resumption). | From ATI start (visit Phase C week 32) to cART resumption up to week 56
  Proportion of participants who develop new mutations not present in the pre-cART genotype conferring clinically-significant resistance to antiretroviral drugs (out of the individuals not reaching viral re-suppression 12 weeks after cART resumption).
Proportion of participants who suppress pVL to <50 copies/mL 12 weeks after cART resumption. | 12 weeks after cART resumption.
  Proportion of participants who suppress pVL to <50 copies/mL 12 weeks after cART resumption.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Mothe, MD, PhD, Principal Investigator — IrsiCaixa AIDS Research Institute, Hospital Universitari Germans Trias i Pujol
Locations (1):
- IrsiCaixa AIDS Research Institute, Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bailon L, Llano A, Cedeno S, Escriba T, Rosas-Umbert M, Parera M, Casadella M, Lopez M, Perez F, Oriol-Tordera B, Ruiz-Riol M, Coll J, Perez F, Rivero A, Leselbaum AR, McGowan I, Sengupta D, Wee EG, Hanke T, Paredes R, Alarcon-Soto Y, Clotet B, Noguera-Julian M, Brander C, Molto J, Mothe B; AELIX002 Study Group. Safety, immunogenicity and effect on viral rebound of HTI vaccines in early treated HIV-1 infection: a randomized, placebo-controlled phase 1 trial. Nat Med. 2022 Dec;28(12):2611-2621. doi: 10.1038/s41591-022-02060-2. Epub 2022 Oct 27. PMID 36302893